CLINICAL TRIAL: NCT03277560
Title: MaTOMS: A Feasibility Study Into the Validity and Acceptability of Routine Collection of Outcome Data in Major Trauma Patients in a Major Trauma Centre in England
Brief Title: MaTOMS: A Feasibility Study Into Collecting Major Trauma Outcomes
Acronym: MaTOMS
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Liz Tutton, Senior Research Fellow, Oxford University Hospitals NHS Trust
Other Study IDs: 12/SC/0628
Record Dates: First submitted 2015-01-21; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Trauma
Keywords: Major Trauma Centre; ISS; Outcome Measures
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No Intervention as it is an observational study — No Intervention as it is an observational study

SUMMARY:
Major Trauma Outcome Measures Study (MaTOMS): A feasibility Study into using outcome measures in major trauma patients.

At present patients who suffer major trauma (multiple, serious injuries that could result in death or serious disability e.g. serious head injuries and multiple fractures), are now able to survive due to advances in modern medicine. Unfortunately they may be left with long term disabilities such as problems with performing day to day activities. We currently do not know how bad these disabilities are or have any way of judging any differences between the outcomes of different hospitals.

MaTOMS is a feasibility study taking place in one hospital, the John Radcliffe Hospital which aims to help answer these questions by developing a set of structured interviews that can be used after an injury to find out about patient outcomes. It will identify how difficult or easy it is to collect the data and information outlined in this project, and whether the types of data and information collected as part of the interviews are a good indicator of a patient's outcomes.

Over 30 months the study will recruit up to 100 patients who are aged 2 years and over who have been admitted following major trauma. Major trauma will be defined as a score of 9 or more on the Injury Severity Score, a widely used system to stratify those who suffer an injury.

Those who agree to take part following a consent process will undergo structured interviews both in hospital and twice via telephone in the year following discharge. Some participants will take part in an additional interview either asking about their experience of answering the questions during the structured interview or exploring their experience and feelings about their traumatic injury to see if our structured interviews are missing any aspect of their experience.

The main objectives for this feasibility study is to test the feasibility of routine collection of outcome measurement data following major trauma.

DETAILED DESCRIPTION:
Purpose and design

Historically much of the literature into major trauma refers to outcomes and mortality synonymously. However there is a growing recognition that as trauma systems mature and more patients lives are saved, the focus has to shift from amenable mortality to improving patient morbidity. Other than mortality it is not currently possible to ascertain the outcomes of patients with major trauma in England as there is no international consensus on which outcome measures should be collected for major trauma patients, nor a collection process in place.

Patients who suffer major trauma are often left with significant long term morbidity with one paper suggesting 42% are unable to return to work at 1 year and another suggesting full recovery is only present in 30% at 5 years. It is important for patients and the public that any outcome measures that are implemented can allow the identification of good or inadequate treatment so that attention can be addressed to improving the quality of care. None of these exist at present and this feasibility study aims to help identify and develop these for possible national implementation.

The study is designed as an observational feasibility study as the way outcomes will be assessed is via a structured interview either face to face or by telephone made up of questions from existing outcome measure instruments and the practicalities of collection of data and identification of the best instruments need to be made prior to any larger study. The instruments have been chosen from those that are known to measure outcomes in one or more domains of the World Health Organisation International Classification of Functioning, Disability and Health (WHO ICF) and that have been previously used to measure outcome in major trauma patients in the literature and have been recommended by a workshop of clinicians and other stakeholders.

The study is designed as an observational feasibility study as the way outcomes will be assessed is via a structured interview either face to face or by telephone made up of questions from existing outcome measure instruments and the practicalities of collection of data and identification of the best instruments need to be made prior to any larger study. The instruments have been chosen from those that are known to measure outcomes in one or more domains of the World Health Organisation International Classification of Functioning, Disability and Health (WHO ICF) and that have been previously used to measure outcome in major trauma patients in the literature and have been recommended by a workshop of clinicians and other stakeholders.

The design of the study has been influenced by existing protocols by which major trauma patients are routinely followed up in Victoria State in Australia. The main difference is that whilst the Australian protocols involved optout consent, this study will involve informed consent or in the case of those who are unable to consent, their Consultee (either personal or nominated) will be asked to advise whether they think the patient would be content to participate. Children aged 2 or more will be included in this study with their parents providing informed consent.

This study will build on the current literature as it will allow the assessment of the feasibility of assessing outcomes in an English Major Trauma Centre and the identification of the most suitable instruments. The study will also measure each instruments and their validity & sensitivity to change and allow an estimation of the costs and other logistics surrounding the routine collection of this data in England to be made.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 2 years
* First admission (for a particular set of injuries) to the Major Trauma Centre
* Traumatic injuries with ISS 9 or more as estimated at time of eligibility assessment
* Within 4 weeks of injury

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:
* Non resident in the United Kingdom
* Patient unwilling to give informed consent
* Patient unable to give informed consent and 'consultee' advises they feel patient would not be content to participate
* Inmate in prison and therefore unable to be easily followed up by telephone

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 2 or over who are admitted to the study centre with a diagnosis that is encompassed by the definition of major trauma (Injury Severity Score greater than or equal to 9) following injury will be eligible for the study as long as they are enrolled less than 4 weeks following the injury and consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
EQ-5D | 12 months
  Quality of life

SECONDARY OUTCOMES:
SF12 | 12 months
  Quality of Life
GOS-E | 12 months
  Function
FIM | 12 months
  Function
Pain Score | 12 months
  Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Keith Willett, Principal Investigator — Oxford University Hospital Trust
Locations (1):
- Oxford University Hospital Trust, Oxford, United Kingdom